CLINICAL TRIAL: NCT01427153
Title: Orthopaedic Manual Physical Therapy Versus Corticosteroid Injections for Osteoarthritis of the Knee
Brief Title: A Comparison of Manual Physical Therapy and Corticosteroid Injections for Knee Osteoarthritis
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Madigan Army Medical Center (U.S. Federal Agency)
Collaborators: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dan Rhon, Staff Physical Therapist, Madigan Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 211081
Record Dates: First submitted 2011-08-30; First posted 2011-09-01 (Estimated); Last update posted 2025-01-27 (Actual); Status verified 2020-07

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; physical therapy; corticosteroid; treatment
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Corticosteroid (Active Comparator): Corticosteroid injection
  Interventions: Procedure: Corticosteroid Injection
- Orthopaedic Manual Physical Therapy (Active Comparator): OMPT consists of joint and soft-tissue mobilizations and the exercises that reinforce the manual techniques.
  Interventions: Procedure: Orthopaedic manual physical therapy

INTERVENTIONS:
Procedure: Orthopaedic manual physical therapy — OMPT consists of joint and soft-tissue mobilizations and the exercises that reinforce the manual techniques.
  Arms: Orthopaedic Manual Physical Therapy
Procedure: Corticosteroid Injection — Corticosteroid injection to the tibiofemoral joint
  Arms: Corticosteroid

SUMMARY:
The purpose of this study is to compare an orthopaedic manual physical therapy (OMPT) approach to a corticosteroid injection approach for the management of knee osteoarthritis.

DETAILED DESCRIPTION:
The purpose of this study is to compare a commonly offered clinical approach of a series of intra-articular steroid injections to an orthopaedic manual physical therapy (OMPT) approach consisting of manually applied passive movement and reinforcing exercise for the treatment of osteoarthritis of the knee (knee OA). A second purpose is to validate a clinical prediction rule (CPR) for patients unlikely to respond to the orthopaedic manual physical therapy approach in a pre-planned secondary analysis of data from the randomized clinical trial.

Aim 1: To see if there is a significant difference in pain and function lasting out to 1 year for patients that receive a clinical approach consisting of a series of intra-articular steroid injections compared to those that receive a clinical approach consisting of orthopaedic manual physical therapy.

Aim 2: To validate a clinical prediction rule of characteristics identified in a previous preliminary study that predicted which patients with knee OA would be unlikely to respond to OMPT.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must be eligible for care in the military health system
* Meet Altman's clinical criteria for knee OA
* Have English language skills sufficient to complete the WOMAC and GROC outcome instruments
* Be 38 years of age or older

Exclusion Criteria:

* Steroid injections or physical therapy treatment for their knee in the past 12 months
* Current or past history of rheumatoid arthritis or similar rheumatic condition
* Current or past history of gout or pseudogout of the knee
* Active infection in the knee within the past 12 months
* Other physical ailment or condition that is typically more limiting or painful than their knee OA during activities such as sitting, standing, walking, or stair climbing
* History of allergy or adverse effect to corticosteroids
* Cannot speak/read English adequately to understand and provide consent to participate in the study
* Pregnant or intending to become pregnant
* Military service members pending a medical evaluation board, physical evaluation board, equivalent discharge process, or on medical hold to determine long-term disposition. For non-military personnel, anyone that is pending or undergoing any litigation for this condition.
* Contraindication to receiving a corticosteroid injection (history of allergic or adverse reaction to steroid injection, history of multiple corticosteroid injections in that area even if not within last year, etc)
* Unable to give informed consent to participate in the study.

Min Age: 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Western Ontario McMasters Osteoarthritis Index (WOMAC) | 1 year
  The WOMAC is a self report questionnaire that asks patient to rate their pain, stiffness, and functional limitation associated with their condition. This instrument will provide important information about the self-reported pain and disability level of the patients in this study. The WOMAC is a recommended primary outcome measure in therapy trials of arthritic conditions, and is considered one of the most appropriate scales for trials evaluating knee osteoarthritis (OA). It is a reliable, valid, and responsive instrument widely used in clinical trials evaluating therapy for hip and knee OA

SECONDARY OUTCOMES:
Global Rating of Change (GROC) | 1 Year
  The GROC questionnaire is a common, feasible, and useful method for assessing short term outcomes and overall changes in quality of life, and is a valid measurement of change in patient status in a variety of pain populations. The GROC has a 15-point scale with a change of positive three points or higher demonstrating clinically significant improvement in a patients perception of quality of life.
Alternate Step Test (AST) | 1 Year
  The Alternate Step Test is an inexpensive and efficient measure of dynamic postural stability and mobility. The AST requires participants to alternate feet and step 8 times (4 times for each foot) onto a 18 cm stool or step as rapidly as possible Recent evidence involving community dwelling adults also suggests that the AST has acceptable test-retest reliability (ICC=0.78) and potential as a fall risk assessment measure.
Timed Up and Go Test (TUG) | 1 Year
  The Timed Up and Go Test is a functional performance measure which directly evaluates an individual's ability to transfer, ambulate, and maintain balance during transitions. Individuals are timed on how quickly they can stand, walk 3 meters, turn around, and return to the chair and sit down. The TUG has good inter-rater and intra-rater reliability and validity for functional testing in older adults at risk for falls. The test is easy to administer and can be completed in two to three minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rhon, PT, DPT, DSc, Principal Investigator — Madigan Army Medical Center; Gail Deyle, PT, DPT, DSc, Study Director — Baylor University / Brooke Army Medical Center; Steven Allison, PT, PhD, Study Chair — Baylor University
Locations (2):
- United States (2):
  - Brooke Army Medical Center, San Antonio, Texas
  - Madigan Army Medical Center, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
Any data sharing must go through a Data Sharing Agreement approved by the US Defense Health Agency
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: These are all available in the supplementary appendix published in the trial results with NEJM
Access Criteria: All of this data is publicly available in open access publications and in the supplementary appendix of the version published on NEJM

REFERENCES:
- [Background] Deyle GD, Allison SC, Matekel RL, Ryder MG, Stang JM, Gohdes DD, Hutton JP, Henderson NE, Garber MB. Physical therapy treatment effectiveness for osteoarthritis of the knee: a randomized comparison of supervised clinical exercise and manual therapy procedures versus a home exercise program. Phys Ther. 2005 Dec;85(12):1301-17. PMID 16305269
- [Background] Deyle GD, Henderson NE, Matekel RL, Ryder MG, Garber MB, Allison SC. Effectiveness of manual physical therapy and exercise in osteoarthritis of the knee. A randomized, controlled trial. Ann Intern Med. 2000 Feb 1;132(3):173-81. doi: 10.7326/0003-4819-132-3-200002010-00002. PMID 10651597
- [Background] Hepper CT, Halvorson JJ, Duncan ST, Gregory AJ, Dunn WR, Spindler KP. The efficacy and duration of intra-articular corticosteroid injection for knee osteoarthritis: a systematic review of level I studies. J Am Acad Orthop Surg. 2009 Oct;17(10):638-46. doi: 10.5435/00124635-200910000-00006. PMID 19794221
- [Background] Godwin M, Dawes M. Intra-articular steroid injections for painful knees. Systematic review with meta-analysis. Can Fam Physician. 2004 Feb;50:241-8. PMID 15000335
- [Derived] Rhon DI, Kim M, Asche CV, Allison SC, Allen CS, Deyle GD. Cost-effectiveness of Physical Therapy vs Intra-articular Glucocorticoid Injection for Knee Osteoarthritis: A Secondary Analysis From a Randomized Clinical Trial. JAMA Netw Open. 2022 Jan 4;5(1):e2142709. doi: 10.1001/jamanetworkopen.2021.42709. PMID 35072722
- [Derived] Deyle GD, Allen CS, Allison SC, Gill NW, Hando BR, Petersen EJ, Dusenberry DI, Rhon DI. Physical Therapy versus Glucocorticoid Injection for Osteoarthritis of the Knee. N Engl J Med. 2020 Apr 9;382(15):1420-1429. doi: 10.1056/NEJMoa1905877. PMID 32268027
- [Derived] Deyle GD, Gill NW, Rhon DI, Allen CS, Allison SC, Hando BR, Petersen EJ, Dusenberry DI, Bellamy N. A multicenter randomised, 1-year comparative effectiveness, parallel-group trial protocol of a physical therapy approach compared to corticosteroid injection on pain and function related to knee osteoarthritis (PTA Trial). BMJ Open. 2016 Mar 31;6(3):e010528. doi: 10.1136/bmjopen-2015-010528. PMID 27033961